CLINICAL TRIAL: NCT01502085
Title: A Phase IIb Trial of Vorinostat in Combination With Lenalidomide and Dexamethasone in Multiple Myeloma Patients Refractory to Previous Lenalidomide Containing Regimens
Brief Title: Vorinostat,Lenalinomide and Dexamethasone in Multiple Myeloma Refractory to Previous Lenalinomide Containing Regimens
Acronym: RZD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-2580
Record Dates: First submitted 2011-12-27; First posted 2011-12-30 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat, Lenalinomide, Dexamethasone (Experimental): Vorinostat: 400 mg po days 1-7 and 15-21 Lenalidomide: 25 mg po days 1-21
  * Lenalidomide dose for patients with renal impairment (CrCL<50ml/min) has be dose adjusted according to package insert Dexamethasone: 40mg po days 1, 8, 15 and 22 for patients aged less than 75 years, 20mg for those aged 75 years and above
  Interventions: Drug: Vorinostat, Lenalinomide and Dexamethasone

INTERVENTIONS:
Drug: Vorinostat, Lenalinomide and Dexamethasone — Vorinostat: 400 mg po days 1-7 and 15-21 Lenalidomide: 25 mg po days 1-21
  * Lenalidomide dose for patients with renal impairment (CrCL<50ml/min) has be dose adjusted according to package insert
  Dexamethasone: 40mg po days 1, 8, 15 and 22 for patients aged less than 75 years, 20mg for those aged 75 years and above

SUMMARY:
Phase IIb clinical trial to determine if resistance to a lenalidomide containing regimen can be overcome by the addition of vorinostat, in patients with relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
lenalidomide has been investigated in combination with both lenalidomide and bortezomib regimens. "Investigational" means that the drug is still being studied and that the study doctors are trying to find out more about it; such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating relapsed and/or refractory multiple myeloma.

Lenalidomide is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental because the FDA has not approved this combination. Participants will receive 25mg of lenalidomide on days 1-21 every 28 days.

Vorinostat is a drug that interferes with the life sustaining functions of the tumor cells. It has already received regulatory approval by the U.S. Food and Drug Administration (FDA) for the treatment of T-cell non-Hodgkin's Lymphoma in the United States. The usage of vorinostat in Multiple Myeloma is experimental (investigational) and has not been approved by the FDA, but studies in combination with proteasome inhibitors (bortezomib) and immunomodulatory (lenalidomide) agents are ongoing. Participants will receive either 400mg of vorinostat on days 1-7 and 15-21 every 28 days.

Dexamethasone is a steroid that is known to cause cell death in multiple myeloma. Dexamethasone is FDA approved for the treatment of multiple myeloma and many other disease states. Participants will receive either Dexamethasone 40mg for those less than 75 years of age or 20mg for those aged 75 years and above on days 1, 8, 15 and 22 every 28 days In this research study the investigators are looking to evaluate the safety and efficacy of vorinostat when combined with lenalidomide and dexamethasone in treating relapsed and/or refractory multiple myeloma, refractory to lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible to enroll in this study:

  * International Staging System symptomatic multiple myeloma, as recently defined (Kyle et al., 2009) or Durie-Salmon stage I-III multiple myeloma, after at least one (1) prior anti-myeloma regimen.
  * Refractory to lenalidomide (administered either with dexamethasone or in combination with other agents); refractory will be defined as no response (<MR) or PD on or within 60 days of discontinuing a prior lenalidomide-containing regimen.
  * Measurable monoclonal protein by serum or urine; or FLC level ≥ 10mg/dL (with abnormal FLC ratio), or measurable extramedullary plasmacytomas:
  * No prior HDAC inhibitor
  * Age ≥ 18 years
  * Performance status ECOG 0-3
  * Acceptable organ function as defined by:
* Bilirubin <2 x upper limit of normal
* ALT and AST <2.5 x upper limit of normal
* Serum creatinine <3.0 mg/dL
* ANC ≥1.0 x 109/L
* Platelet count ≥50 x 109/L

  * QTc interval ≤ 470ms
  * Non-pregnant and non-lactating
  * Life expectancy of more than six months
  * Written informed consent in accordance with federal, local and institutional guidelines
  * Females of Child Bearing Potential* (FCBP) must have a negative serum or urine pregnancy test, with a sensitivity of at least 50 mIU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescription must be filled with 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO methods of acceptable methods of birth control, one highly effective method AND one additional effective method of birth control (contraception) AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy Testing. (See Appendix G: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods) *A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
  * Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy (See Appendix G: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods)
  * All study participants must be registered into the mandatory RevAssist® program and be willing and able to comply with the requirements of RevAssist®.
  * Subjects must adhere to the study visit schedule and other protocol requirements and receive outpatient treatment and laboratory monitoring at the institute that administers the drug.
  * Subjects must agree to take enteric-coated aspirin 81-325 mg orally daily, or if history of prior thrombotic disease or allergy to aspirin, must be fully anticoagulated with warfarin (INR 2-3), Pradaxa® or be treated with full-dose, low molecular weight heparin, as if to treat deep venous thrombosis (DVT)/pulmonary embolism.

Exclusion Criteria:

* Subjects must not meet any of the following exclusion criteria to be eligible to enroll in this study:

  * Subjects with non-secretory or hyposecretory multiple myeloma, defined as <0.5 g/dL M-protein in serum and <200 mg/24 hr Bence Jones protein in urine and serum free light chain <10mg/dL (<100 mg/L)
  * Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation
  * Pregnant or breast feeding females
  * CrCl <30 ml/min or renal failure requiring hemodialysis
  * Prior history or malignancy other than multiple myeloma, unless patient has been disease free of the disease for ≥3 years.
  * Prior or local irradiation within two weeks before screening
  * Evidence of central nervous system (CNS) involvement
  * Unable to take corticosteroids at study entry
  * Peripheral neuropathy of ≥ grade 3 severity
  * Inability or unwillingness to comply with birth control requirements
  * Unable to take antithrombotic medicines at study entry
  * Refusal to participate in study
  * Persons protected by a legal regime (guardianship, trusteeship)
  * Chemotherapy with approved or investigative anticancer therapeutics, including steroid therapy dose as defined above, within 3 weeks prior to first dose
  * Congestive heart failure (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction in the previous six months
  * Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
  * Known or suspected HIV infection, known HIV seropositivity, or active hepatitis A, B, or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Siegel, M.D., Ph.D, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat, Lenalinomide, Dexamethasone: Vorinostat: 400 mg po days 1-7 and 15-21 Lenalidomide: 25 mg po days 1-21 * Lenalidomide dose for patients with renal impairment (CrCL<50ml/min) has be dose adjusted according to package insert Dexamethasone: 40mg po days 1, 8, 15 and 22 for patients aged less than 75 years, 20mg for those aged 75 years and above
  Vorinostat, Lenalinomide and Dexamethasone: Vorinostat: 400 mg po days 1-7 and 15-21 Lenalidomide: 25 mg po days 1-21
  * Lenalidomide dose for patients with renal impairment (CrCL<50ml/min) has be dose adjusted according to package insert
  Dexamethasone: 40mg po days 1, 8, 15 and 22 for patients aged less than 75 years, 20mg for those aged 75 years and above
Period: Overall Study
Arm/Group | Vorinostat, Lenalinomide, Dexamethasone
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat, Lenalinomide, Dexamethasone
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (PR or Better) of Vorinostat in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed/Refractory MM Refractory to a Previous Lenalidomide Containing Regimen
Description: Defined as:
  1. Progression on therapy OR within 60 days after the last dose of a lenalidomide containing regimen OR
  2. No clinical response (<MR) on a lenalidomide containing regimen An overall response rate of 25% or more will be acceptable, while an overall response of less than or equal to 16% will be considered unacceptable. Response will be assessed according to a modified International Working Group Uniform Response Criteria (Durie et al., 2006)
     * Complete Response: Negative immunofixation on the serum and urine and Disappearance of any soft tissue plasmacytomas and ⩽5% plasma cells in bone marrow
     * Very Good Partial Response- Serum and urine M-component detectable by immunofixation but not on electrophoresis or 90 or greater reduction in serum M-component plus urine M-component <100 mg per 24 h
     * Partial Response- ⩾50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ⩾90% or to <200 mg per 24 h.
Time Frame: On treatment portion of study is completed after 12 cycles (each cycle is 28 days in duration) and one month of follow up. Patients may be followed for up to two years after last dose of lenalidomide and vorinostat for disease status and survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat, Lenalinomide, Dexamethasone
Number analyzed (Participants) | 25
Participants | 6

ADVERSE EVENTS:
Arm/Group | Vorinostat, Lenalinomide, Dexamethasone
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat, Lenalinomide, Dexamethasone (N=25)
Syncopal Episode (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Viral Syndrome/Neutropenia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat, Lenalinomide, Dexamethasone (N=25)
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Anemia (Blood and lymphatic system disorders) | 13
Fatigue (General disorders) | 18
Diarrhea (Gastrointestinal disorders) | 18
Dysgeusia (Nervous system disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Anorexia (Gastrointestinal disorders) | 7
Hyperglycemia (Blood and lymphatic system disorders) | 5
Abdominal Bloating (Gastrointestinal disorders) | 4
Elevated Liver Function Tests (Hepatobiliary disorders) | 4
Scalp Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Weight Loss (General disorders) | 4
Peripheral Neuropathy (Nervous system disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Abdominal Discomfort (General disorders) | 3
Mood Alteration (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes